CLINICAL TRIAL: NCT05974462
Title: Single-blind, Investigator-initiated, Randomized, Controlled Trial to Assess the Safety and Efficacy of Intravenous Corticosteroid Therapy to Treat Patients With Acute Myocarditis With Mildly Reduced Left Ventricular Ejection Fraction
Brief Title: MYTHS-MR Trial (MYocarditis THerapy With Steroids in Patients With Mildly Reduced Ejection Fraction)
Acronym: MYTHS-MR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-501547-33-00
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Acute Myocarditis
MeSH Terms: interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Single Blind, Investigator-initiated, Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulsed corticosteroid therapy (Experimental): IV methylprednisolone 125 mg daily for 3 days diluted in saline solution 250 ml on top of standard therapy.
  Interventions: Drug: Methylprednisolone 125 MG
- Placebo (Placebo Comparator): IV saline solution 250 mL daily for 3 days on top of standard therapy.
  Interventions: Other: IV saline solution 0.9%

INTERVENTIONS:
Drug: Methylprednisolone 125 MG — 125 mg daily for 3 days diluted in saline solution 250 mL
  Other Names: Solu-Medrol
  Arms: Pulsed corticosteroid therapy
Other: IV saline solution 0.9% — Saline solution 0.9% 250 mL
  Other Names: sodium chloride
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to demonstrate the efficacy of pulsed intravenous methylprednisolone in a single-blind randomized controlled trial versus standard therapy in patients with acute myocarditis and a mildly reduced LVEF.

The main question[s] it aims to answer are:

* is there an increase in LVEF (≥55% or an absolute increase in LVEF ≥ 10%) on echocardiogram after 5 days from randomization in patients treated with pulsed corticosteroid therapy vs. standard therapy?
* is there a reduction in the proportion of patients with LVEF < 55% AND/OR LV dilation on a 6-month CMRI in patients treated pulsed corticosteroid therapy vs. standard therapy?
* To assess the effect of corticosteroids on the occurrence of the combined endpoint(1) all-cause death or (2) HTx or (3) long-term LVAD implant or (4) first rehospitalization due to HF or ventricular arrhythmias, or advanced AV block.

Participants will be randomized in two arms in a 1:1 ratio. The experimental group will receive pulsed corticosteroid therapy on top of the standard therapy and patients in the placebo group will be treated with a saline solution on top of their standard therapy. All other tests are executed according to standard of care.

DETAILED DESCRIPTION:
Acute myocarditis (AM) is a common condition characterized by histological evidence of inflammatory infiltrates associated with myocyte necrosis of non-ischemic origin. Clinical presentation spans from indolent form to cardiogenic shock also called fulminant myocarditis (FM). Patients can be stratified on the basis of their clinical presentation: patients with left ventricular (LV) ejection fraction (EF)<50% at first echocardiogram, and those with sustained ventricular arrhythmias, called complicated AM, have a worse prognosis compared with uncomplicated cases with preserved left ventricular ejection fraction (LVEF) and without arrhythmias. Among complicated AM, FM patients are those ones at the highest risk, presenting with severely impaired LVEF (generally <40%), and with need for inotropes and/or temporary mechanical circulatory supports (t-MCS).The pathogenesis of AM is felt to be due to an immune-mediated response against the myocardium.

As such, the overall objective is to evaluate the efficacy of pulsed IV corticosteroids therapy for the treatment of AM. It is proposed to test the efficacy of pulsed IV methylprednisolone in a single blind randomized controlled trial versus standard therapy on top of maximal support. The rationale for using pulsed corticosteroid therapy in the acute setting (within 3 weeks from cardiac symptoms' onset) to reduce myocardial inflammatory infiltrates favoring recovery appears strong. Nevertheless, no trial has tested this hypothesis in the very acute phase of AM, despite the high mortality rate of this condition and the fact that AM mainly affects young patients.

Currently, no specific medications in the acute phase of lymphocytic AM are recommended beyond supportive therapy with inotropes and t-MCS. One Cochrane review on corticosteroids showed that almost all studies focused on inflammatory cardiomyopathies with 6 months of symptoms of heart failure (HF), and despite an improvement of cardiac function observed in low quality and small size studies, there was no improvement in the survival. In the past, only one study assessed the efficacy of immunosuppression in AM, the Myocarditis Treatment Trial (MTT) that reported no benefit from immunosuppression. Neutral results in the MTT could be ascribed to a delay in the initiation of this potentially effective treatment. Thus, 55% of patients started immunosuppressive therapy after 1 month from the onset of myocarditis, when the left ventricle (LV) was already dilated, as highlighted by a mean LV end-diastolic diameter (EDD) of 64 mm. It is expected that patients with FM have normal LV dimension during the acute phase despite severe LV systolic dysfunction. Based on a study from the current research group, it was observed that FM patients recover most of the LVEF in the first 2 weeks after admission, with a median absolute increase of 30%. This finding further suggests that an immunosuppressive treatment should be started as soon as possible to demonstrate effectiveness. As little has changed in the medical treatment of this condition in the last 30 years, identification of effective drugs is needed.

Patients admitted to hospital for suspected AM complicated by a reduced Left Ventricular Ejection Fraction (LVEF<50%) will be screened for randomization.

Patients will be randomized in the two arms in a 1:1 ratio (Pulsed methylprednisolone therapy vs Placebo). Randomization will be performed with stratification by country.

In the companion MYTHS trial (EudraCT identifier: 2021-000938-34) patients admitted to hospital for suspected AM complicated by acute HF/cardiogenic shock and LV systolic dysfunction will be randomized in a 1:1 ratio (pulsed methylprednisolone therapy vs Placebo).

The primary objective is to demonstrate a reduction in the rate of the primary composite endpoint on patients treated with pulsed methylprednisolone therapy vs. standard therapy and maximal supportive care.

Endpoints will be analyzed according to the following principles:

* Intention-to-treat (ITT) population
* Per Protocol (PP) population:
* "Safety population"
* A sensitivity analysis will also be performed on the previously defined populations after excluding patients (1) with histological diagnosis of giant cell myocarditis (GCM) or (2) who did not reach the final diagnosis of acute myocarditis based on CMRI or histology.

A pooled analysis of the efficacy and safety endpoints that are present both in the MYTHS and MYTHS-MR will be performed.

Sample size calculation: we plan to recruit a total of 184 patients, and we expect that about 5% of these patients or local physicians will refuse randomization. This would leave a total of 174 randomized patients (87 per arm).

Considering as relevant an increment in the probability to reach the primary endpoint from 45% in the placebo group on top of standard therapy to 70% in the pulsed corticosteroid arm (absolute risk difference of 25%), the planned sample size will allow to achieve a power of 0.90 with a one-sided z-test with continuity correction and an overall type I error of 0,025.

Enrollment will be 36 months. The follow-up will be 2 years with an additional 3 months to lock the database.

In parallel , a registry, called MYOCARDITIS REGISTRY will prospectively recruit all patients with acute myocarditis demonstrated by CMRI or EMB who are not eligible for randomization.

The study is supported by a grant from Fonds Wetenschappelijk Onderzoek (FWO call 2021, application nr G034622N) EuCT identifier: 2022-501547-33-01

ELIGIBILITY:
Inclusion Criteria:

* LVEF<50% and LV-EDD<56 mm (parasternal long-axis view) on echocardiogram;
* Increased troponin (3x URL) at the time of randomization;
* Clinical onset of cardiac symptoms within 3 weeks from randomization;
* Excluded coronary artery disease by coronary angiogram in subjects ≥46 years of age, in case myocarditis is not histologically proven;
* Randomization within 120 hours from hospital admission.
* Endomyocardial biopsy (EMB) is not considered necessary before randomization and performing EMB is based on the decision of the local team.

Exclusion Criteria:

* Known systemic autoimmune disorder or other conditions at the time of randomization where immunosuppression is assumed useful. Patients in whom a systemic autoimmune disorder will be diagnosed during hospitalization will be included in the study if randomized, including patients with a diagnosis of cardiac sarcoidosis or GCM). Both patients included in the corticosteroids-treatment arm or in the placebo-treatment arm can receive the standard immunosuppressive therapy used in the center since the diagnosis;
* Patients already on oral/IV chronic corticosteroid therapy or other chronic immunosuppressive therapies (colchicine or nonsteroidal anti-inflammatory drugs [NSAIDs] are not considered immunosuppressive drugs);
* Contraindication to corticosteroids, including allergies to this medication and its excipients;
* Patients with persistent peripheral eosinophilia (persistent eosinophil count >7% of the leukocytes) or known hypereosinophilic syndrome at the time of randomization. Patients in whom eosinophilic myocarditis will be diagnosed on EMB will be included in the study if already randomized. Both patients included in the corticosteroids-treatment arm or in the placebo-treatment arm can receive the standard immunosuppressive therapy used in the center since the diagnosis;
* Myocarditis associated with the ongoing administration of anti-cancer immune checkpoint inhibitor (ICI) agents;
* Previously known chronic cardiac (i.e., previous cardiomyopathy, that does NOT include previous myocarditis if there is a functional recovery at the time of screening);
* Evidence of active bacterial or fungal infectious disease (presence of fever or increased C-reactive protein are not considered exclusion criteria), or suspected bacterial/fungal infection associated with increased levels of procalcitonin (cut-off >10 ng/mL), if the laboratory exam is available in the center;
* Known chronic infective disease, such as HIV infection or tuberculosis;
* Out-of-hospital cardiac arrest;
* Echocardiographic presence of images suggestive of other cardiac diseases (i.e. endocarditis)
* Participants involved in another clinical trial;
* Pregnant women (known pregnancy) or POSITIVE human chorionic gonadotropin (HCG) test measures (urine/blood) for women of 18-50 years of age.
* Any other significant disease with expected life expectancy <12 months (i.e., evidence of irreversible severe brain injury) or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* If LVEF<41%, an N-terminal pro-B-type natriuretic peptide (NT-proBNP) concentration of 1600 pg/mL or more or a B-type natriuretic peptide (BNP) concentration of 400 pg/mL or more; (if LVEF 41%-<50% any NT-proBNP or BNP concentration is allowed).

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | Day 5
  LVEF ≥55% or an absolute increase in LVEF≥10% on echocardiogram after 5 days from randomization (echocardiographic clips will be centrally reviewed in a blind fashion by readers).

SECONDARY OUTCOMES:
Improvement of the composite endpoint | 6 months
  Proportion of patients with LVEF<55% AND/OR LV dilation on 6-month cardiac magnetic resonance imaging (CMRI) (CMRI clips will be centrally reviewed in a blind fashion by readers)
Composite endpoint defined as the time from randomization to the first event | Within 6 months and 2 years
  among: (1) all-cause death or (2) HTx or (3) long-term LVAD implant or (4) first rehospitalization due to HF or ventricular arrhythmias, or advanced AV block.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Van de Heyning, Principal Investigator — University Hospital, Antwerp; Enrico Ammirati, Study Chair — Niguarda Hospital Milano; Nicole Sturkenboom, Study Chair — University Hospital, Antwerp
Locations (19):
- Belgium (5):
  - Antwerp University Hospital, Edegem, Antwerp
  - Onze-Lieve-Vrouwziekenhuis (OLV ziekenhuis), Aalst
  - Middelheim Ziekenhuis, Antwerp
  - Jessa ziekenhuis, Hasselt
  - Universitair ziekenhuis Leuven, Leuven
- Italy (12):
  - Niguarda Hospital, Milan, Milan
  - Azienda USL Toscane SUD Est, Arezzo
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - ASST Spedali Civili di Brescia, Brescia
  - Careggi University Hospital, Florence
  - Alessandro Manzoni hospital, Lecco
  - San Raffaele Hospital, Milan
  - Ospedale Maggiore di Milano, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Toscana Gabriele Monasterio, Pisa
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine
- University Medical Centre of Ljubljana, Ljubljana, Slovenia
- Hospital Universitario A Coruña (CHUAC), A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ammirati E, Frigerio M, Adler ED, Basso C, Birnie DH, Brambatti M, Friedrich MG, Klingel K, Lehtonen J, Moslehi JJ, Pedrotti P, Rimoldi OE, Schultheiss HP, Tschope C, Cooper LT Jr, Camici PG. Management of Acute Myocarditis and Chronic Inflammatory Cardiomyopathy: An Expert Consensus Document. Circ Heart Fail. 2020 Nov;13(11):e007405. doi: 10.1161/CIRCHEARTFAILURE.120.007405. Epub 2020 Nov 12. PMID 33176455
- [Background] Basso C. Myocarditis. N Engl J Med. 2022 Oct 20;387(16):1488-1500. doi: 10.1056/NEJMra2114478. No abstract available. PMID 36260793
- [Background] Kociol RD, Cooper LT, Fang JC, Moslehi JJ, Pang PS, Sabe MA, Shah RV, Sims DB, Thiene G, Vardeny O; American Heart Association Heart Failure and Transplantation Committee of the Council on Clinical Cardiology. Recognition and Initial Management of Fulminant Myocarditis: A Scientific Statement From the American Heart Association. Circulation. 2020 Feb 11;141(6):e69-e92. doi: 10.1161/CIR.0000000000000745. Epub 2020 Jan 6. PMID 31902242
- [Background] Ammirati E, Cipriani M, Moro C, Raineri C, Pini D, Sormani P, Mantovani R, Varrenti M, Pedrotti P, Conca C, Mafrici A, Grosu A, Briguglia D, Guglielmetto S, Perego GB, Colombo S, Caico SI, Giannattasio C, Maestroni A, Carubelli V, Metra M, Lombardi C, Campodonico J, Agostoni P, Peretto G, Scelsi L, Turco A, Di Tano G, Campana C, Belloni A, Morandi F, Mortara A, Ciro A, Senni M, Gavazzi A, Frigerio M, Oliva F, Camici PG; Registro Lombardo delle Miocarditi. Clinical Presentation and Outcome in a Contemporary Cohort of Patients With Acute Myocarditis: Multicenter Lombardy Registry. Circulation. 2018 Sep 11;138(11):1088-1099. doi: 10.1161/CIRCULATIONAHA.118.035319. PMID 29764898
- [Background] Ammirati E, Veronese G, Brambatti M, Merlo M, Cipriani M, Potena L, Sormani P, Aoki T, Sugimura K, Sawamura A, Okumura T, Pinney S, Hong K, Shah P, Braun O, Van de Heyning CM, Montero S, Petrella D, Huang F, Schmidt M, Raineri C, Lala A, Varrenti M, Foa A, Leone O, Gentile P, Artico J, Agostini V, Patel R, Garascia A, Van Craenenbroeck EM, Hirose K, Isotani A, Murohara T, Arita Y, Sionis A, Fabris E, Hashem S, Garcia-Hernando V, Oliva F, Greenberg B, Shimokawa H, Sinagra G, Adler ED, Frigerio M, Camici PG. Fulminant Versus Acute Nonfulminant Myocarditis in Patients With Left Ventricular Systolic Dysfunction. J Am Coll Cardiol. 2019 Jul 23;74(3):299-311. doi: 10.1016/j.jacc.2019.04.063. PMID 31319912
- [Background] Ammirati E, Bizzi E, Veronese G, Groh M, Van de Heyning CM, Lehtonen J, Pineton de Chambrun M, Cereda A, Picchi C, Trotta L, Moslehi JJ, Brucato A. Immunomodulating Therapies in Acute Myocarditis and Recurrent/Acute Pericarditis. Front Med (Lausanne). 2022 Mar 7;9:838564. doi: 10.3389/fmed.2022.838564. eCollection 2022. PMID 35350578
- [Background] Chen HS, Wang W, Wu SN, Liu JP. Corticosteroids for viral myocarditis. Cochrane Database Syst Rev. 2013 Oct 18;2013(10):CD004471. doi: 10.1002/14651858.CD004471.pub3. PMID 24136037
- [Background] Mason JW, O'Connell JB, Herskowitz A, Rose NR, McManus BM, Billingham ME, Moon TE. A clinical trial of immunosuppressive therapy for myocarditis. The Myocarditis Treatment Trial Investigators. N Engl J Med. 1995 Aug 3;333(5):269-75. doi: 10.1056/NEJM199508033330501. PMID 7596370
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A. Corrigendum to: 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC) With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2021 Dec 21;42(48):4901. doi: 10.1093/eurheartj/ehab670. No abstract available. PMID 34649282
- [Background] Ammirati E, Cipriani M, Lilliu M, Sormani P, Varrenti M, Raineri C, Petrella D, Garascia A, Pedrotti P, Roghi A, Bonacina E, Moreo A, Bottiroli M, Gagliardone MP, Mondino M, Ghio S, Totaro R, Turazza FM, Russo CF, Oliva F, Camici PG, Frigerio M. Survival and Left Ventricular Function Changes in Fulminant Versus Nonfulminant Acute Myocarditis. Circulation. 2017 Aug 8;136(6):529-545. doi: 10.1161/CIRCULATIONAHA.117.026386. Epub 2017 Jun 2. PMID 28576783